CLINICAL TRIAL: NCT00597844
Title: Improving Functional Outcomes in Patients With Unilateral Vocal Cord Paralysis: Assessment of Adaptation Using Functional Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-036
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Intrathoracic Malignancies; Unilateral Vocal Cord Paralysis
Keywords: type I thyroplasty; unilateral vocal fold augmentation
MeSH Terms: conditions — Vocal Cord Paralysis

ARMS (2):
- 1 (Experimental): voice evaluation and fMRI prior to surgical rehabilitation of UVCP
  Interventions: Other: voice evaluation and fMRI
- 2 (Other): Healthy volunteers-voice evaluation and fMRI
  Interventions: Other: undergo voice evaluation and fMRI prior

INTERVENTIONS:
Other: voice evaluation and fMRI — will undergo voice evaluation and fMRI prior to surgical rehabilitation of UVCP and in approximately one month and six months following treatment.
  Arms: 1
Other: undergo voice evaluation and fMRI prior — in approximately one month and six months
  Arms: 2

SUMMARY:
The purpose of this study is to see how the brain re-learns to control the larynx in speaking and swallowing when undergoing surgical rehabilitation in the form of either thyroplasty or vocal fold augmentation for unilateral vocal cord paralysis. What is needed is information on how the brain re-learns to control speaking and swallowing so that we can eventually learn how to help patients re-learn faster after their procedure. Functional Magnetic Resonance Imaging (or fMRI) will allow us to image your brain as you speak and swallow. We will produce "brain maps" for speaking, swallowing and hand movements.

DETAILED DESCRIPTION:
The purpose of this investigation is to determine cortical mechanisms of adaptation to surgical rehabilitation of patients with unilateral vocal cord paralysis (UVCP) undergoing either type I thyroplasty or unilateral vocal fold augmentation for the management of unilateral vocal cord paralysis. This study will use the non-invasive imaging technique, Functional Magnetic Resonance Imaging (fMRI), to investigate cortical responses and responses in the larynx of patients with UVCP who have been deemed to be candidates for either type I thyroplasty or unilateral vocal fold augmentation for the purpose of rehabilitating this UVCP. Patterns of brain activity from the fMRI studies will be compared with the preoperative study with each patient serving as their own control for the purpose of evaluating the alterations in sensory motor organization of the brain in response to UVCP. In addition, responses in patients with UVCP will be compared to normal controls. This will allow us to identify the impact on speech and swallowing and the subsequent reorganization which we theorize will occur in response to the vocal cord medialization. Patients will undergo standardized voice evaluation with improvement in voice serving as a secondary endpoint. The results of the current investigation will provide needed information on both central and peripheral mechanisms of adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with UVCP undergoing type I thyroplasty or vocal fold augmentation for rehabilitation of speech and swallowing.
* Inclusion criteria for the healthy subjects:
* From age 18-85

Exclusion Criteria:

* for the UVCP patients includes the following:
* History of significant psychiatric condition (e.g. schizophrenia, obsessive-compulsive disorder, significant dementia),
* History of the following neurological conditions: CVA, seizure disorders, demyelinating conditions, systemic neuromuscular disorders, cerebral palsy, Alzheimer's disease.
* History of previous moderate to severe traumatic brain injury.
* History of significant cardiovascular, gastrointestinal or renal disease (e.g. myocardial infarction within the previous 12 months, significant vaso-occlusive disease, severe or advanced asthma, or renal compromise)
* History of achalasia
* History of dysphagia, odynophagia, or aphasia unrelated to present illness.
* History of significant claustrophobic reactions.
* Standard contraindications to MR examinations (e.g. implanted stimulators, pregnancy).

Exclusion criteria for the healthy subjects includes the following:

* All of the conditions listed for the UVCP patients.
* Significant surgery or previous radiation therapy to the head and neck.
* History of other neoplasms involving the brain, head and neck, or gastrointestinal system.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
utilize fMRI technique to characterize adaptation to alterations in vocal cord morphology, speech & swallowing function in patients with UVCP undergoing procedure for rehab of speech and swallowing, either type I thyroplasty or vocal fold augment. | conclusion of study

SECONDARY OUTCOMES:
is to develop a better understanding of central sensory motor reorganization in a response to both a peripheral injury to the speech and swallowing mechanism and surgical repair of the speech and swallowing mechanism | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Peck, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org